CLINICAL TRIAL: NCT01182805
Title: Radiofrequency-based Speckle Tracking Echocardiography to Evaluate Diastolic Function
Acronym: RF-SPEED
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Pixel Velocity, Inc. / Epsilon Imaging (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Theodore J. Kolias, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RF-SPEED; 5R44HL071379 (NIH)
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study. (Other)
  Interventions: Device: Echocardiography system Ultra DCI Model 5000; Device: Echocardiography machine GE Vivid E9; Device: Diastolic function assessment

INTERVENTIONS:
Device: Echocardiography system Ultra DCI Model 5000 — Each subject will undergo scanning using the investigational echocardiography system (Ultra DCI Model 5000)to measure Diastolic Circumferential Strain Rate during Isovolumic Relaxation (DCSR-IVR) as novel measure of diastolic function.
Device: Echocardiography machine GE Vivid E9 — Each subject will undergo echocardiography using a conventional echocardiography machine to evaluate the early diastolic mitral annular velocity (E-prime) using tissue Doppler as a standard measure of diastolic function.
Device: Diastolic function assessment — Each subject will undergo standard echocardiographic measure of the mitral inflow pattern and invasive catheter-derived measure of left ventricular end-diastolic pressure to determine their diastolic function. This evaluation will be used as the gold standard for this study.

SUMMARY:
The purpose of this study is to evaluate a novel ultrasound system's ability to assess the relaxing properties of the heart compared to current techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a clinically indicated left heart cardiac catheterization will be recruited for the study.

Exclusion Criteria:

* Suspected acute ST elevation myocardial infarction.
* Acute coronary syndrome with active ongoing chest pain
* Known or suspected acute aortic dissection
* Known or suspected cardiac tamponade
* Known history of unoperated constrictive pericarditis
* Known or suspected severe aortic stenosis or severe mitral regurgitation
* Heart rhythm other than sinus rhythm on pre-cath EKG
* Age < 18 years old
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore J Kolias, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All study participants underwent measurement of Diastolic Circumferential Strain Rate during Isovolumic Relaxation as well as measurement of E-prime by tissue Doppler. They also all had evaluation of their diastolic function by the combination of their mitral inflow pattern and invasive measure of left ventricular end-diastolic pressure.
Period: Overall Study
Arm/Group | All Study Participants
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study.
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Circumferential Strain Rate During Isovolumic Relaxation
Description: Diastolic circumferential strain rate during isovolumic relaxation is a novel measure of diastolic function that measures the rate of relaxation of the left ventricle during the interval of isovolumic relaxation (the period of active relaxation). We would expect that a higher value reflects better relaxation, and better diastolic function.
Time Frame: Assessed from echo obtained at time of enrollment
Population: Only 26 subjects had adequate images for assessment of DCSR-IVR and had gold standard assessment of diastolic function, and the analysis was limited to these subjects.
Measure: Mean (Standard Deviation); unit: 1/sec
Groups:
- Normal Diastolic Function: These were the subjects deemed to have normal diastolic function using the gold standard assessment of mitral inflow and LV end-diastolic pressure (E/A 1 - 2 and LVEDP <= 15 mm Hg).
- Grade 1 Diastolic Dysfunction: These were the subjects deemed to have Grade 1 diastolic dysfunction using the gold standard assessment of mitral inflow and LV end-diastolic pressure (E/A < 1.0).
- Grade 2 Diastolic Dysfunction: These were the subjects deemed to have Grade 2 diastolic dysfunction using the gold standard assessment of mitral inflow and LV end-diastolic pressure (E/A 1 - 2 and LVEDP > 15 mm Hg).
Arm/Group | Normal Diastolic Function | Grade 1 Diastolic Dysfunction | Grade 2 Diastolic Dysfunction
Number analyzed (Participants) | 7 | 12 | 7
1/sec | 0.61 (0.21) | 0.37 (0.19) | 0.34 (0.12)

2. Primary Outcome: Early Diastolic Mitral Annular Velocity (E-prime) Using Tissue Doppler
Description: E-prime is a conventional commonly-used parameter of diastolic function. Higher values of E-prime typically reflect better diastolic function.
Time Frame: Assessed from echo obtained at time of enrollment
Population: Only 25 subjects had adequate images for assessment of DCSR-IVR and interpretable tissue Doppler and gold standard assessment of diastolic function, and the analysis was limited to these subjects.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Normal Diastolic Function | Grade 1 Diastolic Dysfunction | Grade 2 Diastolic Dysfunction
Number analyzed (Participants) | 7 | 11 | 7
cm/sec | 8.1 (1.9) | 5.6 (1.7) | 7.0 (1.8)

ADVERSE EVENTS:
Arm/Group | Single Arm Study.
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days